CLINICAL TRIAL: NCT04198883
Title: SINGaporean Program Performed With an eXPANsion Medical Device
Brief Title: SINGaporean Program Performed With an eXPANsion Medical Device (SingXpand)
Acronym: SingXpand
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Because of the Impact of CoviD19 pandemy
Sponsor: CellProthera (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CellProthera
Record Dates: First submitted 2019-07-04; First posted 2019-12-13 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2019-07

CONDITIONS: Heart Attack
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: the design : pilot, single-arm, open-labelled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Protheracytes (Experimental): Single arm study : Stem cells injection called Protheracytes
  Interventions: Combination Product: Protheracytes

INTERVENTIONS:
Combination Product: Protheracytes — Intramyocardiac (LV) injection of stem cells with a dedicated catheter
  Other Names: Biocardia Helix catheter

SUMMARY:
The purpose of the pilot study is to evaluate the safety and the individual efficacy of the use of ProtheraCytes® in patients with acute myocardial infarction and decreased ejection fraction. CD34+ cells will be re-injected using a dedicated catheter pushed through the femoral artery up to the left ventricle, thus avoiding open chest surgery.

DETAILED DESCRIPTION:
Primary Objective : The objective is to establish the safety of the interventional procedure beginning at the first G-CSF administration to 6 months after the injection of autologous expanded CD34+ stem cells (ProtheraCytes®) in AMI patients with a LVEF≤45% after PTCA and stent(s) implantation.

Secondary Objective : The objective is to establish the individual efficacy of the interventional procedure beginning at the first G-CSF administration to 6 months after the injection of autologous expanded CD34+ stem cells (ProtheraCytes®) in AMI patients with a LVEF≤45% after PTCA and stent(s) implantation.

ELIGIBILITY:
Inclusion Criteria:

1. De Novo AMI with or without ST segment elevation and with a detection of rise and/or fall of cardiac biomarker values (troponin) with at least one value above the 99th percentile of the upper reference limit.
2. Anterior wall AMI
3. PTCA and stent(s) implantation (=Day 0)
4. LVEF ≤ 45% after stent(s) implantation: Combination of a LVEF ≤ 45 % and of anterior akinetic segment(s) - by echography at Day 2 ± 1 after stent(s) implantations
5. Age must be ≥ 21 and ≤ 80 years
6. Men and Non-pregnant non-lactating women who take efficacious contraceptive measures such as oral contraceptive medications or efficacious and permanent intra-uterine device (drug eluted or not) (IUD) or subcutaneous permanent contraceptive implants or menopaused women (at least a 2 years confirmed menopause) or surgically sterilized women.
7. Having previously signed a written informed consent prior to any study-specific procedures.
8. LVEF remaining ≤ 45% assessed by a 2nd echography at Day 8 (± 2) after stent(s) implantation.

   If these criteria have been validated, then the following assessments will be carried out only after the 2nd echography
9. LVEF remaining ≤ 45% assessed by cMRI
10. Identification of anterior akinetic segment(s) of interest assessed by cMRI
11. Identification of non-viability of anterior segment(s) of interest assessed by cMRI

Exclusion Criteria:

1. Previous and known symptomatic CHF, from class II to IV (included)
2. History of CABG (Coronary Artery Bypass Surgery) surgery
3. History of former significant mitral valve replacement surgery or heart transplantation.
4. Severe valve disease: mitral, aortic stenosis / insufficiency.
5. Diagnosis of non-ischemic dilated cardiomyopathy due to valvular dysfunction, mitral regurgitation, tachycardia, or myocarditis
6. Aortic stenosis as determined as valve area less than 1 cm2 that prohibits catheter access to LV
7. Presence of a prosthetic / mechanical aortic or mitral valve or heart constrictive device.
8. Documented presence of a known LV thrombus
9. Sepsis
10. Endocarditis
11. Infectious pericarditis
12. Pericardial tamponade
13. Left ventricular aneurysm, collagen tissue disease
14. Severe peripheral vascular disease precluding femoral artery access as determined at the time of original catheterization.
15. Pacemaker, implantable cardiac defibrillator, and intra-cerebral aneurysm clips.
16. History of metallic foreign body in their eye
17. Former or current aortic dissection
18. Inadequate bone marrow function: Haemoglobin < 10 g/dL and Platelet count < 100 x 109 / L
19. Previous G-CSF or other Hematopoietic Growth Factor administrations.
20. Blood transfusion(s) within the previous 4 weeks (to exclude potential non-autologous ACPs (Angiogenic Cells Precursors) in the harvested blood).
21. Hepatic failure or history of liver cirrhosis or hepatic severe impairment.
22. Constitutional or acquired coagulopathy
23. Treated chronic renal failure, or haemodialysis or renal severe impairment (creatinine clearance < 30ml/min).
24. Prior or concomitant malignancies except non-melanoma skin cancer or adequately treated in situ cervical cancer or previous cancer in complete response without any treatment in the last 5 years.
25. History of prior mediastinal radiation exposure
26. Serious underlying medical conditions at the investigator's discretion, which could impair the ability of the patient to participate in the trial (e.g. ongoing infection, active autoimmune disease, Amyotrophic Lateral Sclerosis, Systemic Lupus, Multiple Sclerosis).
27. Chronic immunomodulatory or cytotoxic drug treatment intake.
28. Active bleeding or major surgery within 1 month.
29. Human immunodeficiency HIV1-2, HTLV1, HTLV2
30. History or current Hepatitis B (prior vaccination accepted)
31. History or current Hepatitis C
32. Syphilis
33. Chronic Obstructive Pulmonary Disease.
34. Active participation in any other clinical trials
35. Current or recent treatment (within the 60 days period before PTCA and stent(s) implantation) with another investigational drug or procedure.
36. Any other co-existing conditions that will preclude participation in the study or compromise ability to give informed consent.
37. Requirement of i.v. catecholamines or mechanical hemodynamic support (aortic balloon pump) initiated 24 hours before cMRI.
38. Splenomegaly
39. Phenylketonuria
40. History of iron-Dextran allergy
41. History of murin protein allergy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
MACE,SAE and AE | 1 year
  Description, incidence and assessment of MACE (Major Adverse Cardiac Events), SAE and AE .

SECONDARY OUTCOMES:
Change of Cardiac function assessed by cMRI | 1 year
  Assessment of individual change of cardiac function via cardiac MRI performed at screening, and 3, 6 & 12 months after ProtheraCytes® administration.
  * Assessment of Cardiac Event Free Survival.
  * Median Time assessment between treatment procedure onset and cardiac relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Flandrin, Study Director — CellProthera
Locations (1):
- NHCS, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No